CLINICAL TRIAL: NCT04483882
Title: Utility and Efficacy of Tactile Labeling of Ophthalmic Drops for Identity and Frequency of Administration in Low Vision
Brief Title: Tactile Low Vision Labeling of Ophthalmic Drops
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 20-0087
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-04

CONDITIONS: Low Vision Aids
Keywords: Low Vision, Labeling, Tactile
MeSH Terms: conditions — Vision, Low

STUDY DESIGN:
Intervention Model Description: Single Group, Blinded, Sham controlled study
Who Masked: Participant
Masking Description: Subjects will be blinded to product to be provided for visual and tactile definition of label product and type and frequency of prescription.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase I- Visually Obscured Healthy Subjects (Sham Comparator): Tactile label to be evaluated by healthy subjects without visual defect. Subjects in visually obscuring lenses but without peripheral neuropathies or other tactile deficits will evaluate the tactile labeling product for efficacy in drug identity and dosing definition. .
  Interventions: Device: Tactile Labels for Drug identity and dose frequency
- Phase II- Low Vision Over 50 years of age (Active Comparator): Subjects with documented Low Vision of 20/70 or less or visual field less than 20 degrees will be asked to evaluate tactile labeling product for efficacy in drug identity and dosing definition.
  Interventions: Device: Tactile Labels for Drug identity and dose frequency

INTERVENTIONS:
Device: Tactile Labels for Drug identity and dose frequency — The tactile labeling proposed in this protocol is rigid labeling. A ring-clip has an inner diameter of 12.5cm, an outer diameter of 16 cm, and a height of 1.5 cm. The ring is cut at 2 cm to form a semi-circle allowing it to be clipped onto the bottleneck. The ring clip fits most if not all prescription eye drop bottles. The individual protrusions with shapes at the end can be cut off by the pharmacist to match the frequency of administration prescribed.

SUMMARY:
The purpose of this study is an evaluation of a tactile labeling strategy developed in the Ophthalmology Clinical Research Center at University of Texas Medical Branch (UTMB) in collaboration with the UTMB Maker Space to improve low vision patients capability to identify their topical ophthalmic drop treatments and the frequency with which they should be administered. The labeling strategy includes protrusions as frequency markers and shapes to differentiate between treatments of similar frequency prescription.

DETAILED DESCRIPTION:
The purpose of this study is an evaluation of a tactile labeling strategy developed in the Ophthalmology Clinical Research Center at University of Texas Medical Branch (UTMB) in collaboration with the UTMB Maker Space to improve low vision patients capability to identify their topical ophthalmic drop treatments and the frequency with which they should be administered. The labeling strategy includes protrusions as frequency markers and shapes to differentiate between treatments of similar frequency prescription.

The first aim is to evaluate the patient capability to identify the number of protrusions and therefore the frequency of administration prescribed. This should be completed in a timeframe that is not frustrating or problematic to the patient in practice.

The second aim is to evaluate the patient ability to differentiate between drugs with similar frequencies based on a shape on the frequency protrusions in a tactile manner. This also should be completed in a timeframe that is not over burdensome or frustrating to the patient. The protocol is designed to evaluate this tactile labeling design in the population it is designed to support.

ELIGIBILITY:
IInclusion Criteria:

Phase I:

* Candidates will be healthy adults between 18 and 100 years of age
* Candidates will complete the consent briefing and consent documents prior to participating in any study activities.
* Phase II:Inclusion Criteria:
* Candidates will be between 50 and 100 years of age.
* Candidates will have a BCVA equal to or less than 20/70 or have central vision field less than 20 degrees.
* Candidates will complete the consent briefing and consent documents prior to participating in any study activities.

Exclusion Criteria:

Phase I:

* Candidates who do not complete the consent briefing and indicate consent through completion of consent documents with or without a witness (as indicated by their ability to read the documents for themselves out loud with whatever optical assistance necessary (large print, magnification, optical correction, etc.), prior to any study activity, will not be included in this study.
* History of prior non-compliance or the presence or history of psychiatric condition (including drug or alcohol addiction) that would, in the opinion of the investigator, make it difficult for the subject to comply with the study procedures or follow the investigators instructions.

Phase II;

* Candidates under 50 years or older than 100 years of age will be excluded.
* Candidates with a BCVA better than 20/70 or have central vision field greater than 20 degrees, will be excluded.
* Candidates with comorbidities that in the opinion of the investigator confound their ability to complete the assessments in this study (ie. Advanced neuropathy of the hands, dementia, or mental incapacity) will be excluded.
* Candidates who do not complete the consent briefing and indicate consent through completion of consent documents with or without a witness (as indicated by their ability to read the documents for themselves out loud with whatever optical assistance necessary (large print, magnification, optical correction, etc.), prior to any study activity, will not be included in this study.
* History of prior non-compliance or the presence or history of psychiatric condition (including drug or alcohol addiction) that would, in the opinion of the investigator, make it difficult for the subject to comply with the study procedures or follow the investigators instructions.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Correct Drug Identity by Shape | 2 minutes
  Subjects Assessment and Report of drug identity by shape of label protrusions
Correct Drug Identity by Color | 2 minutes
  Subject Assessment and Report of drug identity by color of tactile label
Correct Dose Frequency by Tactile Protrusions | 2 minutes
  Subject Assessment and Report of Drug Dosing frequency by number of protrusions of tactile label

CONTACTS AND LOCATIONS:
Overall Officials: Praveena Gupta, O.D., Ph.D., Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Ophthalmology Clinical Research Center, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Individual's data will not be shared in an identifiable format.